CLINICAL TRIAL: NCT00433433
Title: The H10 EORTC/GELA/IIL Randomized Intergroup Trial on Early FDG-PET Scan Guided Treatment Adaptation Versus Standard Combined Modality Treatment in Patients With Supradiaphragmatic Stage I/II Hodgkin's Lymphoma
Brief Title: Fludeoxyglucose F 18 PET Scan-Guided Therapy or Standard Therapy in Treating Patients With Previously Untreated Stage I or Stage II Hodgkin's Lymphoma
Acronym: H10
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Collaborators: Lymphoma Study Association (Other); Fondazione Italiana Linfomi - ETS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EORTC-20051; EORTC-20051; GELA-H10; IIL-EORTC-20051; EUDRACT-2005-002765-37; EU-20657
Record Dates: First submitted 2007-02-08; First posted 2007-02-12 (Estimated); Last update posted 2021-02-03 (Actual); Status verified 2021-02

CONDITIONS: Lymphoma
Keywords: adult mixed cellularity Hodgkin lymphoma; adult nodular sclerosis Hodgkin lymphoma; stage I adult Hodgkin lymphoma; stage II adult Hodgkin lymphoma; adult lymphocyte depletion Hodgkin lymphoma
MeSH Terms: conditions — Lymphoma; Hodgkin Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Favorable - Standard - any PET outcome (Active Comparator): ABVDx3 cycles + Involved node RT (IN-RT) 30 Gy (+boost of 6Gy to residual lesions); FDG-PET after two cycles of ABVD for comparison with the experimental arm will be performed but no treatment adaptation will take place.
  Interventions: Drug: ABVD q4 weeks; Radiation: IN-RT 30 Gy (+ boost 6 Gy residual); Procedure: FDG-PET scan
- Favorable - Experimental - PET negative (Experimental): ABVDx2 cycles; then FDG-PET evaluation:
  PET negative: ABVDx2 without further RT (total of 4 cycles!)
  Interventions: Drug: ABVD q4 weeks; Procedure: FDG-PET scan
- Favorable - Experimental - PET positive (Experimental): ABVDx2 cycles; then FDG-PET evaluation:
  PET positive: presumed poor-risk: switch to escalated BEACOPPx2 + INRT30Gy (+boost 6Gy to residual lesions).
  Interventions: Drug: BEACOPP escalated q3 weeks; Radiation: IN-RT 30 Gy (+ boost 6 Gy residual); Procedure: FDG-PET scan
- Unfavorable - Standard - Any PET outcome (Active Comparator): ABVDx4 cycles + IN-RT 30Gy (+boost 6Gy to residual lesions). FDG-PET after two cycles of ABVD for comparison with the experimental arm will be performed but no treatment adaptation will take place.
  Interventions: Drug: ABVD q4 weeks; Radiation: IN-RT 30 Gy (+ boost 6 Gy residual); Procedure: FDG-PET scan
- Unfavorable - Experimental - PET negative (Experimental): ABVDx2 cycles; then FDG-PET evaluation:
  PET negative: ABVDx 4 cycles, without RT (total of 6 cycles)
  Interventions: Drug: ABVD q4 weeks; Procedure: FDG-PET scan
- Unfavorable - Experimental - PET positive (Experimental): ABVDx2 cycles; then FDG-PET evaluation:
  PET positive: presumed poor-risk: switch to escalated BEACOPPx2 + INRT 30Gy (+boost 6Gy to residual lesions).
  Interventions: Drug: BEACOPP escalated q3 weeks; Radiation: IN-RT 30 Gy (+ boost 6 Gy residual); Procedure: FDG-PET scan

INTERVENTIONS:
Drug: ABVD q4 weeks — Doxorubicin 25 mg/m2 i.v. day 1 and 15; Bleomycin 10 mg/m2 i.v./i.m. day 1 and 15; Vinblastine 6 mg/m2 i.v. day 1 and 15; Dacarbazine 375 mg/m2 i.v. day 1 and 15
  Arms: Favorable - Experimental - PET negative; Favorable - Standard - any PET outcome; Unfavorable - Experimental - PET negative; Unfavorable - Standard - Any PET outcome
Drug: BEACOPP escalated q3 weeks — Cyclophosphamide 1250 mg/m2 i.v. day 1; Doxorubicin 35 mg/m2 i.v. day 1; Vincristine 1.4 mg/m2 i.v.(max.2mg) day 8; Bleomycin 10 mg/m2 i.v./i.m. day 8; Etoposide 200 mg/m2/ i.v. day 1 to 3; Procarbazine 100 mg/m2 orally day 1 to 7; Prednisone 40 mg/m2 orally day 1 to 14; G-CSF 5 mcg/kg s.c. day 9 to recovery leukocytes>1.0x109/l
  Arms: Favorable - Experimental - PET positive; Unfavorable - Experimental - PET positive
Radiation: IN-RT 30 Gy (+ boost 6 Gy residual)
  Other Names: Involved-Note Radiation Therapy
  Arms: Favorable - Experimental - PET positive; Favorable - Standard - any PET outcome; Unfavorable - Experimental - PET positive; Unfavorable - Standard - Any PET outcome
Procedure: FDG-PET scan
  Other Names: F-18 fluorodeoxyglucose positron emission tomography scan

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more cancer cells. Diagnostic procedures, such as fludeoxyglucose F 18 positron emission tomography (FDG-PET scan), may help doctors predict a patient's response to treatment and help plan the best treatment. It is not yet known whether FDG-PET scan-guided therapy is more effective than standard therapy in treating Hodgkin's lymphoma.

PURPOSE: This randomized phase III trial is studying FDG-PET scan-guided therapy to see how well it works compared with standard therapy in treating patients with previously untreated stage I or stage II Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Evaluate whether chemotherapy alone is as effective, but less toxic, as combined modality treatment, in terms of progression-free survival (PFS), in patients with favorable or unfavorable supradiaphragmatic stage I or II Hodgkin's lymphoma who are fludeoxglucose F 18 positron emission tomography (FDG-PET) scan negative after two courses of doxorubicin hydrochloride, bleomycin, vinblastine, and dacarbazine (ABVD).

Secondary

* Evaluate whether early change of chemotherapy from ABVD to escalated cyclophosphamide, doxorubicin hydrochloride, vincristine, bleomycin, etoposide, procarbazine hydrochloride, and prednisone (escalated BEACOPP) improves the PFS of patients who are FDG-PET scan positive after two courses of ABVD.
* Confirm that early response by FDG-PET scan is predictive of the outcome of patients randomized to the standard treatment arm.

OUTLINE: This is a multicenter, randomized study. Patients are stratified according to disease prognostic profile (favorable vs unfavorable), participating center, Ann Arbor clinical stage (I vs II), and availability of a baseline fludeoxyglucose F 18 positron emission tomography (FDG-PET) scan (yes vs no). Patients are randomized to 1 of 2 treatment arms.

* Arm I (standard [closed to accrual as of 6/24/2011]): Patients receive ABVD chemotherapy comprising doxorubicin hydrochloride IV, bleomycin IV or intramuscularly (IM), vinblastine IV, and dacarbazine IV on days 1 and 15. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity. Patients with favorable prognostic profile receive 3 courses of ABVD. Patients with unfavorable prognostic profile receive 4 courses of ABVD. Patients undergo FDG-PET scan after completion of 2 courses of ABVD. Beginning 3-4 weeks after completion of ABVD, patients undergo involved-node radiotherapy (INRT) 5 days a week for 4-6 weeks.
* Arm II (experimental): Patients receive ABVD as in arm I for 2 courses and then undergo FDG-PET scan. Further treatment is adapted according to FDG-PET scan result.

  * FDG-PET negative: Patients with favorable prognostic profile receive 1 additional courses of ABVD. Patients with unfavorable prognostic profile receive 2 additional courses of ABVD. Patients with favorable or unfavorable prognostic profiles randomized on or after August 9th 2010 who are FDG-PET negative after two courses of ABVD will receive standard combined modality treatment consisting of ABVD and INRT as in arm I.
  * FDG-PET positive: Patients receive ABVD as in arm I for 2 courses or intensification to escalated BEACOPP chemotherapy comprising cyclophosphamide IV and doxorubicin hydrochloride IV on day 1, vincristine IV and bleomycin IV or IM on day 8, etoposide IV on days 1-3, oral procarbazine hydrochloride on days 1-7, oral prednisone on days 1-14, and filgrastim (G-CSF) subcutaneously beginning on day 9 and continuing until blood count recover. Treatment repeats every 21 days for 2 courses in the absence of disease progression or unacceptable toxicity. Beginning 3-4 weeks after completion of ABVD or BEACOPP, patients undergo INRT 5 days a week for 4-6 weeks.

After completion of study treatment, patients are followed periodically for at least 10 years.

PROJECTED ACCRUAL: A total of 1,797 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed Hodgkin's lymphoma

  * No nodular lymphocyte-predominant subtype (nodular paragranuloma)
* Supradiaphragmatic Ann Arbor clinical stage I or II disease
* Must meet criteria for 1 of the following prognostic subsets:

  * Unfavorable subset, defined as meeting 1 of the following criteria:

    * Clinical stage II disease with ≥ 4 nodal areas involved

      * Mediastinum and hili are considered as 1 nodal area
    * Age ≥ 50 years
    * Erythrocyte sedimentation rate (ESR) ≥ 50 mm/hr with no B symptoms
    * ESR ≥ 30 mm/hr with B symptoms
    * Mediastinum/thoracic (MT) ratio ≥ 0.35
  * Favorable subset, defined as meeting all of the following criteria:

    * Clinical stage I disease OR stage II disease with ≤ 3 involved areas
    * Age < 50 years
    * ESR < 50 mm/hr (no B symptoms) OR ESR < 30 mm/hr (B symptoms present)
    * MT ratio < 0.35
* Previously untreated disease
* Planning to undergo fludeoxyglucose F 18 positron emission tomography after the first 2 courses of study chemotherapy

PATIENT CHARACTERISTICS:

* WHO performance status 0-3
* Bilirubin ≤ 2.5 times upper limit of normal (ULN)
* Creatinine ≤ 2.5 times ULN
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No severe cardiac, pulmonary, neurologic, psychiatric, or metabolic disease
* No unstable diabetes mellitus
* No other malignancies within the past 5 years except for basal cell skin cancer or adequately treated carcinoma in situ of the cervix
* No known HIV infection
* No psychological, familial, sociological, or geographical condition that would preclude study compliance

PRIOR CONCURRENT THERAPY:

* Not specified

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1952 (Actual)
Dates: Start 2006-10 (Actual); Primary Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Progression-free survival

SECONDARY OUTCOMES:
Event-free survival
Overall survival
Long-term toxicity, in terms of secondary malignancies, cardiovascular events, and pulmonary events

CONTACTS AND LOCATIONS:
Overall Officials: John Raemaekers, MD, PhD, Principal Investigator — EORTC - Universitair Medisch Centrum St. Radboud, Nijmegen, NL; H. Eghbali, MD, Study Chair — EORTC - Institut Bergonie, Bordeaux, FR; Marc Andre, MD, Principal Investigator — GELA - Centre Hospitalier Notre Dame - Reine Fabiola, Brussels, BE; Oumedaly Reman, MD, Study Chair — GELA - CHU de Caen, Caen, FR; Massimo Federico, MD, Principal Investigator — GIMEMA- Azienda Ospedaliera - Universitaria di Modena, Modena, IT; Ercole Brusamolino, MD, Principal Investigator — GIMEMA - Fondazione I.R.C.C.S. Policlinico San Matteo, Pavia, IT
Locations (1):
- Universitair Medisch Centrum St. Radboud - Nijmegen, Nijmegen, Netherlands

REFERENCES:
- [Result] André M, Reman O, Fédérico M, et al.: First report on the H10 EORTC/GELA/IIL randomized intergroup trial on early FDG-PET scan guided treatment adaptation versus standard combined modality treatment in patients with supra-diaphragmatic stage I/II Hodgkin's lymphoma, for the Groupe d'Etude Des Lymphomes De l'Adulte (GELA), European Organisation for the Research and Treatment of Cancer (EORTC) Lymphoma Group and the Intergruppo Italiano Linfomi (IIL) . [Abstract] Blood 114 (22): A-97, 2009.
- [Derived] Kreuzberger N, Goldkuhle M, von Tresckow B, Kobe C, Sickinger MT, Monsef I, Skoetz N. Positron emission tomography-adapted therapy for first-line treatment in adults with Hodgkin lymphoma. Cochrane Database Syst Rev. 2025 Mar 26;3(3):CD010533. doi: 10.1002/14651858.CD010533.pub3. PMID 40135712
- [Derived] Phillips EH, Counsell N, Illidge T, Andre M, Aurer I, Fiaccadori V, Fortpied C, Neven A, Federico M, Barrington SF, Raemaekers J, Radford J. Maximum tumor diameter is associated with relapse risk in limited-stage Hodgkin lymphoma: an international study. Blood Adv. 2025 May 13;9(9):2266-2274. doi: 10.1182/bloodadvances.2024015140. PMID 39774828
- [Derived] Fiaccadori V, Neven A, Fortpied C, Aurer I, Andre M, Federico M, Counsell N, Phillips EH, Clifton-Hadley L, Barrington SF, Illidge T, Radford J, Raemaekers JMM. Relapse patterns in early-PET negative, limited-stage Hodgkin lymphoma (HL) after ABVD with or without radiotherapy-a joint analysis of EORTC/LYSA/FIL H10 and NCRI RAPID trials. Br J Haematol. 2023 Mar;200(6):731-739. doi: 10.1111/bjh.18594. Epub 2022 Dec 21. PMID 36541117
- [Derived] Cottereau AS, Versari A, Loft A, Casasnovas O, Bellei M, Ricci R, Bardet S, Castagnoli A, Brice P, Raemaekers J, Deau B, Fortpied C, Raveloarivahy T, Van Zele E, Chartier L, Vander Borght T, Federico M, Hutchings M, Ricardi U, Andre M, Meignan M. Prognostic value of baseline metabolic tumor volume in early-stage Hodgkin lymphoma in the standard arm of the H10 trial. Blood. 2018 Mar 29;131(13):1456-1463. doi: 10.1182/blood-2017-07-795476. Epub 2018 Feb 1. PMID 29437590
- [Derived] Raemaekers JM, Andre MP, Federico M, Girinsky T, Oumedaly R, Brusamolino E, Brice P, Ferme C, van der Maazen R, Gotti M, Bouabdallah R, Sebban CJ, Lievens Y, Re A, Stamatoullas A, Morschhauser F, Lugtenburg PJ, Abruzzese E, Olivier P, Casasnovas RO, van Imhoff G, Raveloarivahy T, Bellei M, van der Borght T, Bardet S, Versari A, Hutchings M, Meignan M, Fortpied C. Omitting radiotherapy in early positron emission tomography-negative stage I/II Hodgkin lymphoma is associated with an increased risk of early relapse: Clinical results of the preplanned interim analysis of the randomized EORTC/LYSA/FIL H10 trial. J Clin Oncol. 2014 Apr 20;32(12):1188-94. doi: 10.1200/JCO.2013.51.9298. Epub 2014 Mar 17. PMID 24637998